CLINICAL TRIAL: NCT02107300
Title: NeutraSal in the Management of Xerostomia in Obstructive Sleep Apnea Syndrome (OSAS) Patients Utilizing Continuous Positive Airway Pressure (CPAP) Therapy
Brief Title: NeutraSal Treatment for Xerostomia in OSAS Patients Using CPAP Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Invado Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CPAP
Record Dates: First submitted 2014-03-28; First posted 2014-04-08 (Estimated); Results first posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Xerostomia
Keywords: Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Xerostomia; Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NeutraSal (Experimental): NeutraSal, dosed 2 times per day at waking and bedtime (indications 2-10 times per day or PRN), swish and spit, daily for a term of 12 weeks.
  Interventions: Drug: NeutraSal
- Placebo (Placebo Comparator): Placebo dosed 2 times per day at waking and bedtime (indications 2-10 times per day or PRN), swish and spit, daily for a term of 12 weeks.
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: NeutraSal — NeutraSal is a powder that when dissolved in water creates a supersaturated calcium phosphate rinse.
  Arms: NeutraSal
Drug: Placebo Comparator — Placebo is a powder consisting of sodium chloride only; chosen to mimic NeutraSal
  Arms: Placebo

SUMMARY:
To assess whether the daily use of NeutraSal will prevent or reduce dry mouth in patients undergoing CPAP therapy for OSAS and improve CPAP compliance

DETAILED DESCRIPTION:
Subjects diagnosed with Obstructive Sleep Apnea Syndrome (OSAS) who have started CPAP treatment and have complained of dry mouth or developed worsening of a pre-existing dry mouth as an effect of CPAP treatment will test the effectiveness of NeutraSal mouthwash in preventing or reducing his/her dry mouth perceptions and improving their compliance with CPAP.

ELIGIBILITY:
Inclusion Criteria:

* Patient should be above 18 years of age.
* Patients who have been initiated on CPAP therapy after an initial diagnosis of OSAS and have developed dry mouth or have worsening of pre-existing dry mouth condition, as an effect of CPAP therapy.
* Ability to attend visits at the research site
* Patient should be able to read and/or understand and sign the consent form be willing to participate in the research study

Exclusion Criteria:

* Patients with open mouth sores at study entry.
* Any pathology that, based on the judgement of the researcher, could negatively affect the oral mucosa and subsequent treatment for xerostomia (immune disorders, etc.)
* Patients using any other prophylactic mouthwashes.
* Patients who are pregnant and/or nursing.
* Patients becoming pregnant during the treatment period will be removed from data.
* Patients on a low sodium diet
* Patients currently on medication or treatment for xerostomia
* Patients < 18 years of age
* Hypersensitivity to any of the following ingredients- sodium chloride, sodium phosphate, calcium chloride and sodium bicarbonate

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-11; Primary Completion 2015-04-10 (Actual); Study Completion 2017-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chitra Lal, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NeutraSal | Placebo
Started | 16 | 15
Completed | 16 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NeutraSal | Placebo | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Full Range); unit: years] | 53.5 [27 to 80] | 54 [37 to 71] | 53.5 [27 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 16 | 15 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 16 | 15 | 31
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31
Overall Number of Baseline Participants [Count of Participants; unit: Participants] | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage of Time With CPAP (Continuous Positive Airway Pressure) Usage
Description: To observe the impact of NeutraSal on OSAS (obstructive sleep apnoea syndrome) patients compliance to CPAP (Continuous Positive Airway Pressure) therapy compared to placebo. CPAP usage is determined by % of nights CPAP use was greater than 4 hours.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | NeutraSal | Placebo
Number analyzed (Participants) | 16 | 15
percentage of time | -5.09 (.27) | 11.67 (.16)

2. Secondary Outcome: Mean Rate of Dry Mouth as Assessed by Xerostomia Questionnaire
Description: To assess whether the daily use of NeutraSal will prevent or reduce dry mouth perception in OSAS patients undergoing CPAP therapy. Dry Mouth perception will be measured by an Xerostomia Questionnaire which rates mouth dryness. The scale is rated from 1-10 (1 being dry as a desert and 10 is normal)
Time Frame: Baseline through 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NeutraSal | Placebo
Number analyzed (Participants) | 16 | 15
score on a scale | .61 (2.78) | .73 (3.33)

ADVERSE EVENTS:
Arm/Group | NeutraSal | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 7/16 | 6/15
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NeutraSal (N=16) | Placebo (N=15)
Neutrasal drug related (General disorders) | 3 (3) | 0 (0) — Reported salty taste, dry mouth because of drug
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
URI (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
URI and aphthoid ulcer (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
URI and sinus infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shingles (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Neck stiffness (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-09-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT02107300/Prot_SAP_000.pdf